CLINICAL TRIAL: NCT07258459
Title: Trial of Labor After Two CS Before and After Training a Protocol Introduction
Brief Title: Two Previous Cesarean and Vaginal Birth Before and After Starting Training and Protocols
Acronym: TOLA2C Train
Status: Recruiting | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Claudio Celentano, MD, G. d'Annunzio University
Other Study IDs: ObGynEASC009
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cesarean Delivery Affecting Fetus or Newborn; Labor (Obstetrics)--Complications; Hemorrhagic Complications
Keywords: previous CS; trial of labor; maternal outcomes; fetal outcomes; neonatal outcomes
MeSH Terms: interventions — Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 2: term pregnant women with 2 previous CS from 01.01.2021 to 31.12.2025
  Interventions: Procedure: Acceptance, rate of vaginal birth and safety
- Group 1: Women with a history of two previous CS in period 01.01.2026 - 31-12.2020
  Interventions: Procedure: Acceptance, rate of vaginal birth and safety

INTERVENTIONS:
Procedure: Acceptance, rate of vaginal birth and safety — In 2021 started a new delivery protocol enhancing the opportunity of having a trial of labor in women with a history of two previous CS. Rate of acceptance, rate of successful vaginal birth, maternal and fetal outcomes were evaluated

SUMMARY:
In 2015 ObGyn Dept of Santo Spirito Hospital in Pescara (Italy) started protocol for previous CS vaginal birth. In 2021 was started a protocol for training on obstetric emergencies and protocol on two previous cesarean was endorsed. Patients attending birth in Pescara with two previous from january 2016 to December 2020, and from january 2021 to december 2025 were collected. A different counseling approach was adopted from 2021. Women's acceptance of trial of labor and maternal and fetal outcomes were collected.

DETAILED DESCRIPTION:
Women attending birth in Santo Spirito Hospital with 2 previous CS were collected.

Exclusion Criteria:

* Patients with clinical indication to CS
* a previous CS less than 18 month before
* breech presentations
* triplets
* premature labor before 34 completed weeks' gestation The first period was starting January 1st 2016 to December 31st 2020. The second period was starting January 1st 2021 to December 31st 2025

Primary outcomes:

* incidence of trial of labor acceptance
* incidence of vaginal birth

Secondary outcomes:

* maternal adverse outcomes (PPH, blood transfusion, vaginal tears, hysterectomy, maternal death)
* fetal adverse outcomes (fetal death, NICU stay, APGAR score less than 7 at 5')

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* pregnancy above 34 weeks' gestation
* cephalic presentation of the fetus
* singleton and twins
* diamniotic twins
* 2 previous CS
* more than 18 months from last CS
* no other indication to CS

Exclusion Criteria:

* pregnancy below 34 weeks' gestation
* breech baby
* triplets or high order multiple pregnancies
* more than 2 previous CS
* less than 18 months from last CS
* precence of other indications to CS (i.e. maternal diseases, placenta previa, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: pregnant women attending birth in Santo Spirito Hospital Pescara (Italy) from 01-01-2016 to 31-12-2025
Sampling Method: Non-Probability Sample
Enrollment: 2016 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
vaginal birth after 2 cesarean | 5 years
  Incidence of patients having a vaginal birth after 2 CS
accepted indication to trial of labor | 5 years
  incidence of women accepting indication to trial of labor

SECONDARY OUTCOMES:
emergency CS | 5 years
  incidence of emergency CS
maternal outcomes | 5 years
  incidence of adverse maternal outcomes (PPH, blood transfusion, vaginal tears, hysterectomy)
Fetal and Neonatal adverse outcomes | 5 years
  Incidence of fetal/neonatal death, NICU stay, APGAR score below 7 at 5'

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Claudio Celentano, Pescara, PE
  - Santo Spirito Hospital, Pescara, PE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brandstetter M, Brandstetter A, Kainz-Schultes S, Jacobs VR, Fazelnia C, Fischer T, Bogner G. Successful Trial of Labor After Two Caesarean Sections (TOLA2C): Analysis of a Delivery Protocol with Feto-Maternal Outcome. Geburtshilfe Frauenheilkd. 2025 Feb 7;85(8):862-869. doi: 10.1055/a-2513-6562. eCollection 2025 Aug. PMID 40771829